CLINICAL TRIAL: NCT01123772
Title: Phase I, Randomized, Double-Masked, Placebo-Controlled, Dose-Escalation Study to Evaluate Tolerability, Safety & PK of BID Topical Ocular Application of INO-8875 in Healthy Older-Adult Volunteers
Brief Title: Phase I Dose-Escalation Study to Evaluate Tolerability, Safety & PK of INO-8875 in Healthy Older-Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Inotek Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IPC-09-2009
Record Dates: First submitted 2010-04-27; First posted 2010-05-14 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Health
Keywords: adenosine agonist; eye drop; elderly volunteer; older healthy volunteer
MeSH Terms: interventions — INO-8875

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (Placebo Comparator): Vehicle control
  Interventions: Other: Placebo control
- INO-8875 (Experimental): Active drug
  Interventions: Drug: INO-8875

INTERVENTIONS:
Drug: INO-8875 — eye drops for 14 days in one eye
  Arms: INO-8875
Other: Placebo control — Matched placebo
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate how tolerable and safe it is to give INO-8875 eye drops at different concentrations to normal older healthy adult volunteers for two weeks.

ELIGIBILITY:
Inclusion Criteria:

* male, or a female with a negative pregnancy test and without childbearing potential
* aged 35 to 65 years
* body weight is ≥50 kg and ≤115 kg

Exclusion Criteria:

* Subject has glaucoma or any active ophthalmologic disease including conjunctivitis
* Subject has a central retinal vein occlusion in either eye at any time in the past
* Subject is currently on any drug that might affect IOP including oral or ocular glucocorticoids or ephedrine
* Subject has history of ocular trauma or surgery (except for non-incisional surgery performed at least 3 months prior to the Screening visit)
* Subject has a prosthetic eye or any ocular abnormality precluding reliable applanation tonometry in either eye including an immobile pupil.
* Subject is not able to refrain from use of contact lenses during the Treatment Period

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2010-05; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Evansville, Indiana, United States